CLINICAL TRIAL: NCT03640546
Title: Program Evaluation of Connections, a Healthy Marriage and Responsible Fatherhood (HMRF) Grant Funded Program.
Brief Title: Healthy Marriage and Responsible Fatherhood Grant Program With Phoenix House of New York
Acronym: HMRF-CP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Phoenix House Foundation, Inc. (Other)
Collaborators: New York University (Other)
Responsible Party: Sponsor
Other Study IDs: 90FM0110-01-00
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Relationship, Family; Substance Use; Parenting
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Within My Reach/ Within Our Reach — Relationship education workshops

SUMMARY:
The purpose of this study is to provide a process and outcome evaluation of the HMRF grant-funded Connections program. Phoenix Houses of New York, Inc. has been given a new grant to continue and refine its successful Connections program which equips single and coupled participants with significant substance use disorders (SUD) with the skills and knowledge needed to (1) create and/or sustain healthy relationships/marriages, (2) equip participants with the skills and knowledge to raise children in a functional and healthy environment, (3) improve their financial stability, job readiness and employability to improve economic self-sufficiency and responsibility, and (4) reduce relationship stress and strain on interactions between co-parents.

DETAILED DESCRIPTION:
The process evaluation will focus on:

* Documenting project implementations and determining efficient replication methods for effective program components,
* Monitoring completion of overall program goals and objectives, and
* Allow for quality improvement during the five year grant cycle.

The outcome evaluation which focuses on participant level impact will ask the following:

* Does participation in evidence-based relationship education improve healthy relationship skills for single or coupled enrollees?
* Does participation in partner education and support classes improve co-parenting relationship?
* Do participants have better attitudes toward their ability to manage money (i.e. savings, paying bills) after workshops in financial literacy and other money management services?
* Do participants have improved attitudes on their own employability after workshops targeted at job readiness?
* Does participation in job readiness preparation translate into improved employment prospects or readiness factors? (Readiness factors may include increased family assets and economic status.)
* Does participation in family care management sessions improve marriage/relationship, child and family well-being?
* Does participation in parenting education improve parenting skills and attitudes toward parenting? Does participation in parenting education improve commitment to parenting and children?

ELIGIBILITY:
Inclusion Criteria:

* Adult Phoenix House clients who are enrolled in Connections evidence-based interventions

Exclusion Criteria:

* Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults in romantic relationships with or without children
Sampling Method: Non-Probability Sample
Enrollment: 3825 (Estimated)
Dates: Start 2016-05-27 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Healthy Relationship Skills | 0 days, 30 days, and 90 days
  Evidence-based curriculum scale. Questionnaire Items range on a scale from (1) Strongly Disagree to (5) Strongly Agree. Generally a higher response indicates a better outcome however some items are reverse-coded.

SECONDARY OUTCOMES:
Change in co-parenting relationship and attitudes towards parenting | 0 days and 90 days
  Parenting curriculum scale. Questionnaire Items range on a scale from (1) Strongly Disagree to (4) Strongly Agree. Generally a higher response indicates a better outcome however some items are reverse-coded.
Change in job readiness and attitudes towards employability | 0 days and 90 days
  Vocational Scale. Questions are on a yes or no scale, with yes indicating a better response.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Phoenix House - Hauppauge, Hauppauge, New York
  - Phoenix House - Long Island City, Long Island City, New York
  - Phoenix House - Ronkonkoma, Ronkonkoma, New York

IPD SHARING:
Plan to Share IPD: No